CLINICAL TRIAL: NCT03219229
Title: Metabolic Effects of Differential Organ Growth Rates
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Dympna Gallagher, Professor of Nutritional Medicine, Columbia University
Other Study IDs: AAAO3053
Record Dates: First submitted 2017-07-11; First posted 2017-07-17 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Resting Energy Expenditure
Keywords: Fat-free mass; Tanner stage 1; Pre-pubertal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prepubertal children: Healthy 7-11 year old girls and boys.

SUMMARY:
Young children have a high resting energy expenditure (REE) relative to their body weight and metabolically active compartment, fat-free mass (FFM). Both body weight and FFM are, however, metabolically heterogeneous and include organs and tissues varying widely in specific metabolic rate (i.e., organ REE/kg/d). One prevailing hypothesis is that most, if not all, of the higher REE observed in young animals and children compared to adults can be accounted for by a larger proportion of high metabolic rate components such as brain, liver, and heart..

DETAILED DESCRIPTION:
FFM was the traditional and only means of adjusting REE for between-individual differences in metabolically active tissue components. The investigators seek to improve the understanding of variation in REE by developing new and improved rapid magnetic resonance imaging (MRI) methods of quantifying some of the major heat producing organs and tissues in children and adults. The long-term aim is to provide an improved understanding of human energy requirements. Specifically, the investigators propose to test whether: 1) a portion of the elevated daily REE adjusted for FFM observed in young children (Tanner Stage 1) could be accounted for by the relative fractions of body mass as high metabolic activity tissues (heart, liver, kidney, brain) and low metabolic activity tissues (skeletal muscle, adipose tissue), 2) a portion of the age-related decline in daily REE adjusted for FFM observed in children could be accounted for by changes in the relative fractions of body mass as high and low metabolic rate tissues during growth.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Aged from 7-11 years
* Pre-pubertal (based on Tanner staging)
* Africa-American, Asian, and Caucasian (by self-report of all 4 grandparents of same race group)

Exclusion Criteria:

* Actively involved in a weight management program
* Have co-morbidities of obesity (Blounts disease, hypertension, diabetes; sleep apnea)
* Have entered puberty
* Precocious puberty
* Have known metabolic abnormalities
* Were born prematurely, or were small or large for gestational age
* Lean individuals who have a family history (parents or siblings) of obesity or Type 2 diabetes
* Current or previous significant use of any medication known to affect any of the variables being measured

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects will be healthy African-American, Asian (Chinese, Korean, Japanese), and Caucasian pre-pubertal females and males (ages 7-11 years) at baseline. Lean (Body mass index (BMI) < 85th by age and sex) and obese (BMI > 95th percentile by age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2004-02-14 (Actual); Primary Completion 2007-02-20 (Actual); Study Completion 2007-02-20 (Actual)

PRIMARY OUTCOMES:
Resting energy expenditure in kilocalories | Day 1
  REE is measured by indirect calorimetry over a 30 minute period and extrapolated to a 24 hour period
Fat mass in kilograms | Day 1
  Measured from a whole-body dual energy X-ray absorptiometry (DXA) scan
Fat-free mass in kilograms | Day 1
  Measured from a whole-body dual energy X-ray absorptiometry (DXA) scan
Height in meters | Day 1
  Measured using a stadiometer
Weight in kilograms | Day 1
  Measured using a calibrated scale
Liver in kilograms | Day 1
  Total volume measured by MRI
Heart in kilogram | Day 1
  Left ventricular mass measured by cardiac gated MRI
Kidneys in kilogram | Day 1
  Total volume measured by MRI
Spleen in kilograms | Day 1
  Total volume measured by MRI
Trunk high metabolic rate organs in kilograms | Day 1
  The sum of liver, kidneys, spleen, and heart
Brain mass in kilogram | Day 1
  Total volume measured by MRI
Skeletal muscle mass in kilograms | Day 1
  Skeletal muscle volume measured by MRI
Residual fat-free mass in kilograms | Day 1
  Fat-free mass minus the sum of kidneys, liver, spleen, heart, and skeletal muscle
Total body adipose tissue mass in kilogram | Day 1
  Represents the sum of visceral, subcutaneous, and intermuscular adipose tissue by MRI
Body mass index in kg/m2 | Day 1
  Weight and height will be combined to report BMI
Variability in resting energy expenditure | Day 1
  The collected measures will be aggregated to statistically test the following question: How much of the variability in resting energy expenditure can be accounted for by the mass of the measured organs (liver, kidneys, spleen, heart) and tissues (fat, skeletal muscle, brain) and is the explained variance greater than the variance explained when predicting resting energy explained from a model using fat and fat-free mass alone.

SECONDARY OUTCOMES:
Change in resting energy expenditure in relation to changes in body composition and organ mass. | From baseline measure to follow-up, approximately 2 years
  A portion of age-related decline (2-years) in daily REE adjusted for FFM observed in children is explainable in part by changes in the relative fractions of body mass as high (brain, heart, liver, kidney) and low (skeletal muscle, adipose tissue) metabolic activity tissues with growth and pubertal progress

CONTACTS AND LOCATIONS:
Overall Officials: Dympna Gallagher, Principal Investigator — Columbia University
Locations (1):
- Dympna Gallagher, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bauer J, Thornton J, Heymsfield S, Kelly K, Ramirez A, Gidwani S, Gallagher D. Dual-energy X-ray absorptiometry prediction of adipose tissue depots in children and adolescents. Pediatr Res. 2012 Oct;72(4):420-5. doi: 10.1038/pr.2012.100. Epub 2012 Jul 20. PMID 22821057
- [Result] Dorsey KB, Thornton JC, Heymsfield SB, Gallagher D. Greater lean tissue and skeletal muscle mass are associated with higher bone mineral content in children. Nutr Metab (Lond). 2010 May 11;7:41. doi: 10.1186/1743-7075-7-41. PMID 20459832
- [Result] Shen W, Velasquez G, Chen J, Jin Y, Heymsfield SB, Gallagher D, Pi-Sunyer FX. Comparison of the relationship between bone marrow adipose tissue and volumetric bone mineral density in children and adults. J Clin Densitom. 2014 Jan-Mar;17(1):163-9. doi: 10.1016/j.jocd.2013.02.009. Epub 2013 Mar 21. PMID 23522982
- [Result] Gao Y, Zong K, Gao Z, Rubin MR, Chen J, Heymsfield SB, Gallagher D, Shen W. Magnetic resonance imaging-measured bone marrow adipose tissue area is inversely related to cortical bone area in children and adolescents aged 5-18 years. J Clin Densitom. 2015 Apr-Jun;18(2):203-8. doi: 10.1016/j.jocd.2015.03.002. Epub 2015 Apr 1. PMID 25840474